CLINICAL TRIAL: NCT00932880
Title: An Open-Label, Randomized, Two-Way Crossover, Single Dose Study to Evaluate the Bioavailability of the Test Formulation of Amlodipine 10 mg Tablets [Torrent Pharmaceuticals Limited,India] Compared to a 10 mg Dose of Norvasc®, [Pfizer, USA] in 18 Fed, Healthy Adult Subjects
Brief Title: Study to Evaluate the Bioavailability of the Test Formulation of Amlodipine 10 mg Tablets (Torrent Pharmaceuticals Limited) Compared to a 10 mg Dose of Norvasc® (Pfizer) in 18 Fed, Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Torrent Pharmaceuticals Limited (Industry)
Other Study IDs: 20-061-SA
Record Dates: First submitted 2009-07-01; First posted 2009-07-03 (Estimated); Last update posted 2009-07-16 (Estimated); Status verified 2009-07

CONDITIONS: Healthy
MeSH Terms: interventions — Amlodipine

INTERVENTIONS:
Drug: Amlodipine Besylate — 10 mg tablets (Torrent Pharmaceuticals, India)
Drug: Norvasc — 10 mg dose (Pfizer, USA)

SUMMARY:
* Objective:

  * The objective of this study was to compare the rate and extent of absorption of the test formulation, amlodipine besylate 10 mg tablets (Torrent Pharmaceuticals Ltd.), with that of the marketed reference product, Norvasc® 10 mg tablets (Pfizer, Inc.), when administered under fed conditions.
* Study Design:

  * This was an open-label, randomized, two-way crossover study in which 18 healthy subjects were scheduled to receive a single dose of each of two treatments in two assigned dosing periods. Each dose administration was separated by a minimum 14-day washout period.

ELIGIBILITY:
Inclusion Criteria:

* Sex: Male/female.
* Age: 18 - 45 years.
* Volunteer with BMI of 18-27 kg/m2 with minimum of 50 kg weight.
* With minimum blood pressure of 110/75 mmHg.
* Healthy and willing to participate in the study.
* Signed Written Informed Consent for Screening and study.
* Medical case history, physical examination, vital signs, laboratory tests and ECG without significant deviations.
* Negative drug of abuse screening test.
* Non-smokers or smoking less than 10 cigarettes a day and willing to break smoking in the course of the study.
* No history of medication for at least 2 weeks prior to study drug administration until study Period II completion.

Exclusion Criteria:

* Clinically relevant abnormal physical findings at the screening examination, which would interfere with the objectives of the study.
* Clinically relevant abnormalities in the results of the laboratory screening evaluation.
* Abnormal ECG.
* Habituation of tobacco necessitating uninterrupted tobacco consumption.
* Addiction to alcohol or history of any drug abuse.
* History of kidney or liver dysfunction.
* History of allergy to the test drug or any drug chemically similar to the drug under investigation.
* Administration/ Intake of any prescription or OTC medication for two weeks before the study.
* Patients suffering from any chronic illness such as arthritis, asthma etc.
* HIV, HCV, HBsAg positive volunteers.
* Opioids and cannabis positive volunteers based on urine test.
* Subjects suffering from any psychiatric (acute or chronic) illness.
* Administration of any investigational drug in the period 0 to 3 months before entry to the study.
* Intake of barbiturates or any enzyme-inducing drug in last three months.
* History of significant blood loss due to any reason, including blood donation in the past 12 weeks. The total blood loss in last 3 months including for this study will not exceed 350ml.
* History of any bleeding disorder.
* Existence of any surgical or medical condition, which, in the judgement of the clinical investigator, might interfere with the absorption, distribution, metabolism or excretion of the drug or likely to compromise the safety of volunteers.
* Serious adverse reaction or hypersensitivity to study drug or any of the excipients.
* Inability to communicate or co-operate with the investigator due to language problem, poor mental development or impaired cerebral function.
* Pregnant and nursing mother.
* Female not practicing barrier contraceptives.
* Contraindications to active or inactive ingredients of the formulation.
* Volunteers leaving to go on a holiday.
* Imminent reassignment of job location.
* Inadequate motivation.
* Can not come for the follow-up visits.

Ages: 18 Years to 45 Years | Sex: All
Age Groups: Adult

PRIMARY OUTCOMES:
Bioequivalence

CONTACTS AND LOCATIONS:
Locations (1):
- CEDRA Clinical Research, LLC, San Antonio, Texas, United States